CLINICAL TRIAL: NCT00645918
Title: GRAVITAS: Gauging Responsiveness With A VerifyNow Assay-Impact On Thrombosis And Safety
Acronym: GRAVITAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accumetrics, Inc. (Industry)
Responsible Party: Matthew J. Price, M.D., Scripps Advanced Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: P95082
Record Dates: First submitted 2008-03-24; First posted 2008-03-28 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Arteriosclerosis; Acute Coronary Syndrome
Keywords: Platelets; Platelet Function Tests; Clopidogrel; Drug Eluting Stents; Acute Coronary Syndrome; Myocardial Ischemia; Stent Thrombosis; Heart Diseases; Coronary Disease; Arterial Occlusive Disease
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Ischemia; Heart Diseases; Coronary Disease; Arterial Occlusive Diseases | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): "Tailored" clopidogrel regimen - an additional clopidogrel 600-mg loading dose (eight 75-mg tablets taken orally; daily 150 mg clopidogrel dose plus additional 450 mg clopidogrel) on the day of randomization and then 150-mg clopidogrel every day thereafter for 6 months.
  Interventions: Drug: clopidogrel
- B (Placebo Comparator): "Standard" clopidogrel regimen - a placebo loading dose (six placebo tablets taken orally plus daily dose of one placebo tablet plus 75 mg clopidogrel) on the day of randomization followed by one placebo tablet plus 75 mg clopidogrel every day thereafter for 6 months.
  Interventions: Drug: clopidogrel; Drug: placebo
- C (Placebo Comparator): Responders: A random sample of clopidogrel responders treated with a placebo loading dose (six placebo tablets taken orally plus daily dose of one placebo tablet plus 75 mg clopidogrel) on the day of randomization followed by one placebo tablet plus 75 mg clopidogrel every day thereafter for 6 months.
  Interventions: Drug: clopidogrel; Drug: placebo

INTERVENTIONS:
Drug: clopidogrel — oral, 75 mg daily for 6 months starting on day of randomization
Drug: placebo — oral, 6 pill loading dose on day of randomization; one pill daily for 6 months starting on day of randomization
  Arms: B; C
Drug: clopidogrel — oral, 450 mg loading dose on day of randomization; 75 mg daily for 6 months starting on day of randomization
  Arms: A

SUMMARY:
The objective of the GRAVITAS trial is to determine whether tailored anti-platelet therapy using the Accumetrics VerifyNow P2Y12 assay reduces major adverse cardiovascular events after drug-eluting stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older.
* 2. Patients undergoing coronary angiography and possible PCI with planned use of at least one drug-eluting stent (DES), and without planned use of glycoprotein IIb/IIIa inhibitors. One or more bare metal stents (BMS) may be implanted, and other lesions may be treated without stenting, as long as at least one DES is implanted. However, the procedure must be successful and uncomplicated for all lesions (DES + BMS + non stent).
* Indication for the procedure may be stable angina or ischemia, unstable angina, non-ST elevation MI (NSTEMI), or ST elevation MI (STEMI).
* Have the ability to understand the requirements of the study, including consent for use and disclosure of research-related health information.
* Have the ability to comply with study procedures and protocol, including required study visits.
* 6. A female patient is eligible to enter the study if she is (1) of child-bearing potential and not pregnant or nursing; (2) not of child-bearing potential (i.e., has had a hysterectomy, have both ovaries removed, has tubal ligation, or are post-menopausal, defined as 24 months without menses).

Exclusion Criteria: Pre-PCI

* PCI within previous 30 days.
* Prior consent to participate in GRAVITAS and not randomized by IVRS.
* History of gastro-intestinal bleeding within 6 months.
* Major non-cardiac surgery within 6 weeks.
* Ischemic stroke within 6 weeks.
* Any history of hemorrhagic stroke or sub-arachnoid hemorrhage.
* Other bleeding diathesis, or considered by investigator to be at high-risk for bleeding on long-term clopidogrel therapy.
* Minor surgical procedures that require cessation of dual anti platelet therapy and result in significant bleeding are NOT eligible.
* Current or planned therapy with coumadin anticoagulation.
* Current or planned therapy with other thienopyridine class of ADP receptor inhibitors (e.g., prasugrel, ticlopidine), or the non-thienopyridine ticagrelor.
* Severe allergy to stainless steel, contrast dye, unfractionated heparin, low molecular weight heparin, or bivalirudin that cannot be adequately pre-medicated.
* Allergy to aspirin or clopidogrel.
* Current enrollment in an investigational drug or device study that has not reached the time period of the primary endpoint.
* Have received GPIIb/IIIa inhibitors eptifibatide or tirofiban within 24 hours before or during PCI or abciximab within 10 days before or during PCI.
* Thrombocytopenia (defined as platelet count < 100 K).
* Anemia (hematocrit < 30%).
* Polycythemia (hematocrit > 52%).
* Patients unwilling or unable to complete clinical follow-up for the duration of the study.

Exclusion Criteria: Post-PCI

* PCI with placement of at least one DES is not performed.
* Planned staged PCI in the next 6 months post-procedure.
* Unsuccessful PCI (post-procedure diameter stenosis >30% with less than TIMI-3 flow in any treated vessel).
* Patients with in-hospital STEMI confirmed by ECG prior to randomization or those whom require a target vessel revascularization of the index lesion prior to randomization.
* Patients with acute stent thrombosis before Accumetrics VerifyNow tests.
* Administration of any GPIIb/IIIa during PCI procedure or prior to initial hospital discharge.
* Failure to meet clopidogrel requirements
* Major complication during or after PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of post-randomization CV death, non-fatal MI, or ARC definite/probable stent thrombosis in non-responders randomized to standard vs. tailored dosage | 6 months

SECONDARY OUTCOMES:
Time to first occurrence of post-randomization CV death, non-fatal MI, or ARC definite/probable stent thrombosis in non-responders randomized to standard dosage vs. responders | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Price, M.D., Principal Investigator — Scripps Advanced Clnical Trials
Locations (82):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scottsdale Health Care - Osborn Campus, Scottsdale, Arizona
  - Scottsdale Health Care - Shea Campus, Scottsdale, Arizona
  - Scripps Green Hospital, La Jolla, California
  - El Camino Hospital, Mountain View, California
  - UC Davis Medical Center, Sacramento, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - Alvarado Hospital, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - UCSF Moffitt-Long Hospital, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Torrance Memorial Medical Center, Torrance, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Christiana Care Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Cardiology Research Associates, Ormond Beach, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - St. Joseph's Research Institute, Atlanta, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - St. Vincent Heart Center of Indiana/The Care Group LLC, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - The Lahey Clinic, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Joseph's Mercy Hospital, Ypsilanti, Michigan
  - St. Mary's Duluth Clinic Health System, Duluth, Minnesota
  - St. Luke's / Mid America Heart Institute, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Lenox Hill Hospital, New York, New York
  - NY Presbyterian / Weill Cornell Medical Center, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - North Ohio Research, Ltd., Elyria, Ohio
  - Cleveland Cardiovascular Research Foundation, Fairview Park, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - Geisinger Clinic - Cardiology, Danville, Pennsylvania
  - St. Vincent Health Center, Erie, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - South Austin Hospital, Austin, Texas
  - Austin Heart P.A., Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - University Hospital San Antonio (UTHSCSA), San Antonio, Texas
  - Tomball Regional Hospital, Tomball, Texas
- Canada (10):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario
  - York PCI Group, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM) Hôtel-Dieu, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Montréal Heart Institute, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec

REFERENCES:
- [Derived] Price MJ, Angiolillo DJ, Teirstein PS, Lillie E, Manoukian SV, Berger PB, Tanguay JF, Cannon CP, Topol EJ. Platelet reactivity and cardiovascular outcomes after percutaneous coronary intervention: a time-dependent analysis of the Gauging Responsiveness with a VerifyNow P2Y12 assay: Impact on Thrombosis and Safety (GRAVITAS) trial. Circulation. 2011 Sep 6;124(10):1132-7. doi: 10.1161/CIRCULATIONAHA.111.029165. Epub 2011 Aug 29. PMID 21875913
- [Derived] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Derived] Price MJ, Berger PB, Angiolillo DJ, Teirstein PS, Tanguay JF, Kandzari DE, Cannon CP, Topol EJ. Evaluation of individualized clopidogrel therapy after drug-eluting stent implantation in patients with high residual platelet reactivity: design and rationale of the GRAVITAS trial. Am Heart J. 2009 May;157(5):818-24, 824.e1. doi: 10.1016/j.ahj.2009.02.012. PMID 19376306